CLINICAL TRIAL: NCT02615886
Title: Pilot Feasibility of Dietary Heat-Stabilized Rice Bran Supplementation for Diarrheal Disease Prevention in Nicaraguan Children
Brief Title: Pilot Feasibility of Rice Bran Supplementation in Nicaraguan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Autonomous University of Nicaragua (Other); Virginia Polytechnic Institute and State University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Elizabeth P Ryan, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-5233H
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Dietary Rice Bran Supplementation
Keywords: rice bran; infants; stool metabolome; stool microbiome; dietary intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational Control (Experimental): Randomized participants will be observed for diarrhea incidences throughout the 6 month trial with no intervention.
  Interventions: Other: Observational Control
- Rice Bran (Experimental): Randomized participants will consume a measured dose of rice bran daily throughout the 6 month trial.
  Interventions: Dietary Supplement: Rice bran

INTERVENTIONS:
Other: Observational Control — Participants will be observed and not provided any dietary supplementation.
  Arms: Observational Control
Dietary Supplement: Rice bran — Dietary rice bran consumed daily and amounts increase throughout the 6 month intervention (6 months of age: 1 g/day rice bran, 7 months: 2 g/day rice bran, 8 months: 2 g/day, 9 months: 3g/day, 10 months: 4g/day, 11 months: 5g/day).
  Other Names: whole food dietary intervention
  Arms: Rice Bran

SUMMARY:
The purpose is to assess feasibility of rice bran consumption in weaning children and collect pilot data on gut microbiome and metabolome modulation with rice bran intake for diarrheal prevention.

DETAILED DESCRIPTION:
Rice bran is a globally accessible, underutilized food ingredient with an array of beneficial nutrients (e.g. phytochemicals and prebiotics) that promote health and potentially prevent diseases. The investigators will determine if dietary rice bran intake can modulate the infant gut microbiome and metabolome to promote gut immunity for the benefit of preventing diarrheal diseases that increase risk for malnutrition and stunting.

The investigators hope to learn about the feasibility of dietary supplementation of heat-stabilized rice bran in weaning children living in regions with increased susceptibility to diarrhea and malnutrition, and whether or not rice bran consumption can modulate the stool microbiome and metabolome.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4 months and 6 months at beginning of recruitment
* Have received the 3 doses of the rotavirus vaccination (RV5)
* Families willing to feed their infant a daily dose of study-provided heat-stabilized rice bran for 6 months

Exclusion Criteria:

* Have had a diarrheal episode between 4 and 6 months of age
* Have had a prior hospitalization
* Have had an antibiotic or prophylactic treatment within 1 month prior to participation
* Have an ongoing illness, a known immunocompromising condition, or use of medications

Ages: 4 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who are compliant to consuming rice bran daily and in amounts provided | 6 months
  Record daily rice bran consumption and track compliance to diet intervention by regular visits from local study personnel.

SECONDARY OUTCOMES:
Number of participants with microbial modulations in stool as detected by microbiome sequencing. | 6 months
  Measure the stool microbiome modulation with rice bran consumption for gut health and diarrhea prevention compared to no rice bran consumption.
Number of participants with metabolite modulations in stool as detected by Gas Chromatography-Mass Spectrometry (GC-MS) and Liquid Chromatography-Mass Spectrometry (LC-MS) | 6 months
  Measure the stool metabolome modulation with rice bran consumption for gut health and diarrheal prevention compared to no rice bran consumption.

CONTACTS AND LOCATIONS:
Locations (2):
- Colorado State University, Fort Collins, Colorado, United States
- National Autonomous University of Nicaragua, León, León, Nicaragua

REFERENCES:
- [Background] Goodyear A, Kumar A, Ehrhart EJ, Swanson KS, Grusak MA, Leach JE, Dow SW, McClung A, Ryan EP. Dietary rice bran supplementation differentially prevents Salmonella colonization across varieties and by priming intestinal immunity. J Funct Foods. 2015 Oct;18A: 653-64.
- [Background] Yang X, Wen K, Tin C, Li G, Wang H, Kocher J, Pelzer K, Ryan E, Yuan L. Dietary rice bran protects against rotavirus diarrhea and promotes Th1-type immune responses to human rotavirus vaccine in gnotobiotic pigs. Clin Vaccine Immunol. 2014 Oct;21(10):1396-403. doi: 10.1128/CVI.00210-14. Epub 2014 Jul 30. PMID 25080551
- [Background] Borresen EC, Ryan EP. Rice Bran: A food ingredient with Global Public Health Opportunities In: Watson RR, Preedy, V. R. and Zibadi, S.,editor. Wheat and Rice in Disease Prevention and Health: Benefits, risks, and mechanisms of whole grains in health promotion. 1st ed. Oxford, UK: Elsevier; 2014 p. 301-11.
- [Background] Kumar A, Henderson A, Forster GM, Goodyear AW, Weir TL, Leach JE, Dow SW, Ryan EP. Dietary rice bran promotes resistance to Salmonella enterica serovar Typhimurium colonization in mice. BMC Microbiol. 2012 Jul 4;12:71. doi: 10.1186/1471-2180-12-71. PMID 22583915
- [Background] Henderson AJ, Kumar A, Barnett B, Dow SW, Ryan EP. Consumption of rice bran increases mucosal immunoglobulin A concentrations and numbers of intestinal Lactobacillus spp. J Med Food. 2012 May;15(5):469-75. doi: 10.1089/jmf.2011.0213. Epub 2012 Jan 16. PMID 22248178
- [Derived] Zambrana LE, Weber AM, Borresen EC, Zarei I, Perez J, Perez C, Rodriguez I, Becker-Dreps S, Yuan L, Vilchez S, Ryan EP. Daily Rice Bran Consumption for 6 Months Influences Serum Glucagon-Like Peptide 2 and Metabolite Profiles without Differences in Trace Elements and Heavy Metals in Weaning Nicaraguan Infants at 12 Months of Age. Curr Dev Nutr. 2021 Jul 21;5(9):nzab101. doi: 10.1093/cdn/nzab101. eCollection 2021 Sep. PMID 34514286